CLINICAL TRIAL: NCT04521426
Title: Ventilator-associated Injury (VAI) in Chronic Home Mechanical Ventilation: a Paradigm Switch in Order to Improve Ventilatory Support
Brief Title: Ventilator-associated Injury (VAI) in Chronic Home Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marieke Duiverman, Principal Investigator, University Medical Center Groningen
Other Study IDs: VAI-HMV
Record Dates: First submitted 2020-07-29; First posted 2020-08-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Failure; Long-term Non-invasive Ventilation
Keywords: COPD; Lung fibrosis; non-invasive ventilation; respiratory muscles; diaphragm; lung inflammation; ventilator-induced lung injury
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis; Pneumonia; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Blood samples
  2. BAL fluid
  3. Explanted lungs
  4. Respiratory muscle biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lung Fibrosis: 1. probable or confirmed diagnosis of interstitial pulmonary fibrosis (IPF) or other fibrotic lung disease of unknown origin.
  2. being listed for lung transplantation
  Interventions: Other: No other than standard care
- COPD standard therapy: 1. COPD: GOLD stage III or IV
  2. being listed for lung transplantation
  3. did not underwent LVR surgery or endoscopic LVR
  4. not being treated with chronic NIV
  Interventions: Other: No other than standard care
- COPD with long-term NIV: 1. COPD: GOLD stage III or IV
  2. being listed for lung transplantation
  3. did not underwent LVR surgery or endoscopic LVR
  4. being treated with chronic NIV before lung transplantation (at least 1 months, at least 4 hours per day).
  Interventions: Other: No other than standard care

INTERVENTIONS:
Other: No other than standard care — No other than standard care.

SUMMARY:
Rationale:

The pathophysiological changes in respiratory muscle morphology and functioning in patients with end-stage pulmonary disease are not very well known. Furthermore, in COPD, long-term high-intensity NIV is applied without knowing the exact consequences on the lungs and respiratory muscles.

Objective: The aims of the study are to get insight in:

A. changes respiratory muscles in end-stage respiratory disease, comparing COPD with restrictive lung disease (RLD) due to pulmonary fibrosis B. the effects of long-term HI-NIV in severe COPD patients on the respiratory muscles and the lungs; by comparing COPD patients that had been treated with long-term NIV to COPD patients that were not treated with long-term NIV.

Study design: In order to investigate this, the investigators will include in a small pilot cohort study patients being lung transplanted. In these patients there is lung tissue available and respiratory muscle biopsies will be performed during lung-transplant surgery.

Study population: Patients that are listed for lung transplantation for an underlying diagnosis of COPD or RLD will be asked to participate. Three groups will be included: patients with a RLD due to pulmonary fibrosis, COPD patients that had been treated with long-term NIV prior to being lung transplanted and COPD patients that were not treated with long-term NIV. Patients will be included definitely once being lung transplanted.

Main study parameters/endpoints: The study is an exploratory pilot study. Both contractile strength and the structure of single diaphragm and intercostal muscle fibres as well as lung injury; i.e. alveolar structure and damage and inflammation in the alveoli, will be investigated.

DETAILED DESCRIPTION:
Rationale:

Chronic Obstructive Pulmonary Disease (COPD) is a progressive inflammatory disease characterised by airway and lung parenchyma damage. At end-stage disease patients may develop chronic hypercapnic respiratory failure, a disease characteristic that is however not uniformly seen in other end-stage lung diseases, such as in patients with pulmonary fibrosis. The underlying process for the development of chronic hypercapnic respiratory failure is incompletely understood and the role of respiratory muscle alterations is unclear.

Home noninvasive ventilation with high-intensity ventilatory settings (HI-NIV) has been shown to be effective in these severe COPD patients. However, in patients being mechanically ventilated on the intensive care unit for diverse reasons, high-intensity ventilation, especially high tidal volumes, has been shown to result in ventilator associated lung and diaphragm injury. Whether this occurs in home high-intensity NIV, is however completely unknown.

Objective: The aims of the study are to get insight in:

A. changes respiratory muscles in end-stage respiratory disease, comparing COPD with restrictive lung disease (RLD) due to pulmonary fibrosis B. the effects of long-term HI-NIV in severe COPD patients on the respiratory muscles; i.e. the contractile strength and the structure of single diaphragm and intercostal muscle fibres and the lungs; i.e. alveolar structure and damage and inflammation, by comparing COPD patients that had been treated with long-term NIV to COPD patients that were not treated with long-term NIV.

Study design: In order to investigate this, the investigators will include in a small pilot cohort study patients being lung transplanted. In these patients there is lung tissue available and respiratory muscle biopsies will be performed during lung-transplant surgery.

Study population: Patients that are listed for lung transplantation for an underlying diagnosis of COPD or RLD will be asked to participate. Three groups will be included: patients with a RLD due to pulmonary fibrosis, COPD patients that had been treated with long-term NIV prior to being lung transplanted and COPD patients that were not treated with long-term NIV. Patients will be included definitely once being lung transplanted.

Main study parameters/endpoints: The study is an exploratory pilot study. The study aims to get data on respiratory muscle and lung and airway pathology in order to, if important results are observed, set up a larger prospective trial investigating both clinical outcomes and pathology of the respiratory muscles/lungs. Both contractile strength and the structure of single diaphragm and intercostal muscle fibres as well as lung injury; i.e. alveolar structure and damage and inflammation in the alveoli, will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. RLD: probable or confirmed diagnosis of interstitial pulmonary fibrosis (IPF) or other fibrotic lung disease of unknown origin.
2. COPD: GOLD stage III or IV
3. Being listed for lung transplantation

Exclusion Criteria:

1. Concomitant neuromuscular or systemic/collagen-vascular disease
2. Prior lung surgery (except for lung biopsies) or lung volume reduction treatment
3. Being unable to understand the patient information and consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see above
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle morphology and functioning | during surgery
  Biopsies of the diaphragm and intercostal muscles will be taken during surgery
Ventilator-associated lung injury serum TNF-alfa | during surgery
  serum TNF-alfa
Ventilator-associated lung injury serum IL-6 | during surgery
  serum IL-6
Ventilator-associated lung injury serum IL-1beta | during surgery
  serum IL-1beta
Ventilator-associated lung injury serum IL-8 | during surgery
  serum IL-8
Ventilator-associated lung injury serum MIP-2 | during surgery
  serum MIP-2
Ventilator-associated lung injury serum sRAGE | during surgery
  serum sRAGE
Ventilator-associated lung injury BAL TNF-alfa | during surgery
  BAL TNF-alfa
Ventilator-associated lung injury BAL IL-6 | during surgery
  BAL IL-6
Ventilator-associated lung injury BAL IL-1beta | during surgery
  BAL IL-1beta
Ventilator-associated lung injury BAL IL-8 | during surgery
  BAL IL-8
Ventilator-associated lung injury BAL MIP-2 | during surgery
  BAL MIP-2
Ventilator-associated lung injury BAL sRAGE | during surgery
  BAL sRAGE
Ventilator-associated lung injury basal membrane | during surgery
  histopathological changes to the basal membrane
Ventilator-associated lung injury alveolar cells | during surgery
  histopathological changes to type I alveolar cells
Ventilator-associated lung injury edema | during surgery
  edema in the alveoli and interstitium
Ventilator-associated lung injury fibrin | during surgery
  interstitial fibrin
Ventilator-associated lung injury inflammatory cells | during surgery
  Inflammatory cells influx in the alveoli
Ventilator-associated lung injury gene-expression | during surgery
  Gene-expression profiling of epithelial cells with regard to inflammatory factors

SECONDARY OUTCOMES:
Ventilatory use | during surgery
  Duration of usage (longitudinally and use per day)
Ventilatory settings | during surgery
  Settings of the NIV
Demographics_age | during surgery
  age
Demographics_gender | during surgery
  gender
Demographics_BMI | during surgery
  BMI
Lung Function_FEV1 | during surgery
  FEV1
Lung Function_FVC | during surgery
  FVC
Blood gasses_PaCO2 | during surgery
  PaCO2
Blood gasses_HCO3- | during surgery
  HCO3-

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided